CLINICAL TRIAL: NCT01222845
Title: Glycaemic, Insulinaemic and Appetite Responses to Two Different Types of Porridge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Principal Investigator, Javier Gonzalez, PhD Student, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 32W4
Record Dates: First submitted 2010-10-12; First posted 2010-10-18 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-05

CONDITIONS: Postprandial Glycaemia,; Postprandial Insulinaemia; Appetite

ARMS (2):
- Pinhead oat porridge (Experimental)
  Interventions: Drug: Test meal
- Rolled oat porridge (Experimental)
  Interventions: Drug: Test meal

INTERVENTIONS:
Drug: Test meal — Porridge made from rolled, or pinhead oats providing 50 g of carbohydrate

SUMMARY:
The purpose of this study is to assess the postprandial glycaemic, insulinaemic and appetite responses to porridge made with oats processed differently.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Aged 18-40 years

Exclusion Criteria:

* Food allergies
* Metabolic disorders

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2010-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Blood glucose | Measured at baseline, 15, 30, 45, 60, 90 and 120 min after ingestion of a test meal

SECONDARY OUTCOMES:
Plasma insulin | Measured at baseline, 15, 30, 45, 60, 90 and 120 min after ingestion of a test meal
Subjective appetite ratings | Measured at baseline, 15, 30, 45, 60, 90 and 120 min after ingestion of a test meal
  Measured by a visual analogue scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Emma J Stevenson, PhD, Principal Investigator — Northumbria University
Locations (1):
- Brain, Performance and Nutrition Centre, Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

REFERENCES:
- [Derived] Gonzalez JT, Stevenson EJ. Postprandial glycemia and appetite sensations in response to porridge made with rolled and pinhead oats. J Am Coll Nutr. 2012 Apr;31(2):111-6. doi: 10.1080/07315724.2012.10720016. PMID 22855916